CLINICAL TRIAL: NCT00603083
Title: Postoperative Pain Treatment in Total Hip Arthroplasty A Randomized Double-blinded Placebo-controlled Study to Assess the Effect of Local Analgesia
Brief Title: Postoperative Pain Treatment in Total Hip Arthroplasty: A Study to Assess the Effect of Local Analgesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vejle Hospital (Other)
Responsible Party: Principal Investigator, Per Kjaersgaard-Andersen, Per Kjaersgaard-Andersen MD, Vejle Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EudraCT number 2007-003890-20; S-20070066
Record Dates: First submitted 2008-01-02; First posted 2008-01-28 (Estimated); Last update posted 2011-12-09 (Estimated); Status verified 2011-12

CONDITIONS: Pain, Postoperative
Keywords: Hip Arthroplasty; Treatment Outcome; Local Anesthesia
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine; Ketorolac; Epinephrine; Ketorolac Tromethamine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): This group receive local analgesic with Ropivacaine 200 mg, Ketorolac 30 mg and Adrenaline 1 mg 10 and 22 hours after the operation. The medicine solution is given in a catheter, wich is placed in the hip at the end of the operation.
  Interventions: Drug: Ropivacaine, Ketorolac and Adrenalin
- B (Placebo Comparator): This group receive Placebo 10 and 22 hours after the operation. The Placebo is given in a catheter, wich is placed in the hip at the end of the operation.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ropivacaine, Ketorolac and Adrenalin — The local analgesic with Ropivacaine 200 mg, Ketorolac 30 mg and Adrenaline 1 mg is given 10 and 22 hours after the operation. The medicine solution is administrated in a catheter, which is placed in the hip at the end of the operation.
  Other Names: Naropin; Toradol
  Arms: A
Drug: Placebo — This group receive Placebo 10 and 22 hours after the operation. The Placebo is given in a catheter, which is placed in the hip at the end of the operation.
  Other Names: Saline
  Arms: B

SUMMARY:
The purpose of this study is to determine whether the investigator standardized pain treatment plus local pain treatment is more effective than the investigator standardized pain treatment plus placebo in total hip arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for an uncemented unilateral Total Hip Replacement because of osteoarthritis
* Willingness and possibility to follow the instructions of the study
* 18 years or older
* written informed consent and authority after it has been read and understood.

Exclusion Criteria:

* Operation with anterior approach or using navigation
* Do not understand or speech danish
* Can not use the pain-score Numerical Rating Scale (NRS)
* Special indications for Total Hip Replacement
* Anaesthetized in general anaesthesia where a tube is demanded
* Daily use of strong opioids, based on the investigators assessment
* Fertile women
* ASA-score: 3 and 4
* Known allergy against the standardized pain treatment, the study drugs and placebo, Ropivacaine, Ketorolac, Adrenalin.
* Treatment with Lithium, Dihydroergotamin, full anticoagulant treatment or MAO-inhibitor
* Following illness:
* Active gastric ulcer or earlier gastrointestinal bleeding, ulceration or perforation of any kind.
* Suspicions of manifest gastrointestinal bleeding and/or cerebrovascular bleeding
* Haemorrhagic diathesis
* Coagulation disorder
* Severe thrombocytopenia
* Severe heart insufficiency
* Severe risk of postoperative bleeding or delayed haemostatic
* Myocardium hypertrophy or ischaemic heart disease
* Hypertension
* Hypovolemics
* Anhydration
* angiooedema
* Asthma
* Bronchospasm
* Severe liver insufficiency
* Rhinostenosis because of polyostotic
* Narrow-angled glaucoma
* Phaeochromocytoma
* Low plasm-potassium
* Thyreotoxicosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-01; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Pain score | 24 hours
Opioid Consumption | 24 hours

SECONDARY OUTCOMES:
Pain score | 7 days
Opioid consumption | 3 days
Postoperative Nausea and Vomiting (PONV) | 3 days
Fatigue | 3 days
Physical function | 2 month

CONTACTS AND LOCATIONS:
Overall Officials: Per Kjaersgaard-Andersen, MD, Principal Investigator — Ortopaedic Department, Vejle Hospital, Denmark
Locations (2):
- Denmark (2):
  - Orthopaedic Department, Vejle
  - Ortopaedic Department, Vejle Hospital, Vejle